CLINICAL TRIAL: NCT06579989
Title: Usefulness and Feasibility of Ultrasound in Office Laryngology Procedures: A Pilot Study
Brief Title: Usefulness and Feasibility of Ultrasound in Office Laryngology Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-10026663
Record Dates: First submitted 2024-08-19; First posted 2024-08-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cough; Vocal Cord Atrophy; Vocal Cord Paresis; Vocal Cord Paralysis; Dysphagia; Dysphonia
MeSH Terms: conditions — Cough; Vocal Cord Paralysis; Deglutition Disorders; Dysphonia | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cough (Experimental): Adult patients who are seen at the Sean Parker Institute for the Voice and are determined to have neurogenic cough for which superior laryngeal nerve block is recommended will undergo this procedure under ultrasound guidance. Patients without neurogenic cough will also be recruited for ultrasound assessment to establish landmarks and normal variation.
  Interventions: Diagnostic Test: Ultrasound for cough
- Vocal Cord Atrophy (Experimental): Adult patients with vocal fold atrophy, paresis, or paralysis diagnosed at the Sean Parker Institute for the Voice who are planned to undergo injection laryngoplasty will be invited to take part in the study.
  Interventions: Diagnostic Test: Ultrasound for vocal fold atrophy or vocal fold paresis/paralysis
- Vocal Cord Paresis (Experimental): Adult patients with vocal fold atrophy, paresis, or paralysis diagnosed at the Sean Parker Institute for the Voice who are planned to undergo injection laryngoplasty will be invited to take part in the study.
  Interventions: Diagnostic Test: Ultrasound for vocal fold atrophy or vocal fold paresis/paralysis
- Vocal Cord Paralysis (Experimental): Adult patients with vocal fold atrophy, paresis, or paralysis diagnosed at the Sean Parker Institute for the Voice who are planned to undergo injection laryngoplasty will be invited to take part in the study.
  Interventions: Diagnostic Test: Ultrasound for vocal fold atrophy or vocal fold paresis/paralysis
- Dysphagia (Experimental): Adult patients referred to the Sean Parker Institute for the Voice for swallowing assessment will undergo standard medical history including collection of age, gender, occupation, characteristics of swallowing complaints, and prior evaluation and treatments. Adult patients without swallowing complaints will also be recruited to define normal anatomy and variation.
  Interventions: Diagnostic Test: Ultrasound for dysphagia
- Dysphonia (Experimental): Adult patients referred to the Sean Parker Institute for the Voice for voice assessment will undergo standard medical history including collection of age, gender, occupation, characteristics of voice complaints, and prior evaluation and treatments. Additionally, patients diagnosed with muscle tension dysphonia will be evaluated by ultrasound for the presence, size, and function of their suprahyoid musculature.
  Interventions: Diagnostic Test: Ultrasound for dysphonia

INTERVENTIONS:
Diagnostic Test: Ultrasound for cough — Adult patients who are seen at the Sean Parker Institute for the Voice and are determined to have neurogenic cough for which superior laryngeal nerve block is recommended will undergo this procedure under ultrasound guidance. Patients without neurogenic cough will also be recruited for ultrasound assessment to establish landmarks and normal variation. Patients will be assessed for their comfort with undergoing the procedure and clinicians will be surveyed on the ease and benefit of performing the procedure under ultrasound guidance.
  Arms: Cough
Diagnostic Test: Ultrasound for vocal fold atrophy or vocal fold paresis/paralysis — Adult patients who are seen at the Sean Parker Institute for the Voice and are determined to have vocal fold atrophy or vocal fold paresis/paralysis for whom injection laryngoplasty is recommended will undergo laryngeal ultrasound prior to the procedure to assess baseline anatomy as well as following the procedure (both immediately following the procedure as well as at follow-up visits) in order to assess the amount of injectate.
  Arms: Vocal Cord Atrophy; Vocal Cord Paralysis; Vocal Cord Paresis
Diagnostic Test: Ultrasound for dysphagia — Patients with and without swallowing complaints will be enrolled to assess their tongue, suprahyoid and infrahyoid musculature, including muscle identification, bulk and function.
  Arms: Dysphagia
Diagnostic Test: Ultrasound for dysphonia — Adult patients who are seen at the Sean Parker Institute for the Voice and are determined to have muscle tension dysphonia will undergo ultrasonography during their visit with laryngology or speech language pathology.
  Arms: Dysphonia

SUMMARY:
Investigators will assess the usefulness of using ultrasound in office procedures for laryngology interventions. Participants who qualify will be adults who are undergoing superior laryngeal nerve block, injection laryngoplasty, swallowing evaluation, voice evaluation and voice therapy.

ELIGIBILITY:
Inclusion Criteria:

* US-Guided Injection for Neurogenic Cough:

  1. Age over 18 years
  2. Recommended to undergo superior laryngeal nerve block
* US-Assessment of Superior Laryngeal Nerve Anatomy

  1. Age over 18 years
  2. No cough complaints
* US-Assessment of Injectate Volume:

  1. Documentation of unilateral vocal fold paresis/paralysis or atrophy
  2. Age over 18 years
  3. Recommended to undergo injection laryngoplasty
* US-Assessment of Swallow:

  1. Age over 18 years
  2. Presents with swallowing complaints
* US-Assessment of Normal Swallow:

  1. Age over 18 years
  2. Presents without swallowing complaints
* US-Assessment of Voice:

  1. Age over 18 years
  2. Undergoing evaluation of voice problems

Exclusion Criteria:

1. Age under 18 years and over 99 years
2. Open neck wound including tracheostomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative clinician-reported usability measure of ultrasound during injection of the internal branch of superior laryngeal nerve for neurogenic cough. | Immediately post-intervention
  The clinician will use the Likert scale and rate a series of statements on a scale of 1 (strongly disagree) to 5 (strongly agree). The lowest possible total score is 12 (overall clinician disagreement), and the highest possible total score is 60 (overall clinician agreement).
Qualitative clinician-reported usability measure of ultrasound during injection of the internal branch of superior laryngeal nerve for neurogenic cough. | Immediately post-intervention
  The clinician will respond to the following open-ended questions:
  * What are the benefits with performing the procedure with ultrasound?
  * What are the limitations with performing this procedure with ultrasound?
Patient comfort measures during ultrasound-guided injection of the internal branch of superior laryngeal nerve for neurogenic cough. | Day 1
  Number of patients that fall into the below categories as determined by the provider care team:
  * No discomfort: talking/comfortable throughout
  * Minimal discomfort: 1 or 2 episodes of mild discomfort with no distress
  * Mild discomfort: More than 2 episodes of discomfort without distress
  * Moderate discomfort: significant discomfort experienced several times with some distress
  * Severe discomfort: frequent discomfort with significant distress
Time to complete superior laryngeal nerve injection under ultrasound. | Day 1
  The amount of time will be recorded in minutes.
Images and descriptors of internal branch of superior laryngeal nerve anatomy and normal variation. | Day 1
  This is a qualitative outcome measure. Providers will provide a description of the internal branch of superior laryngeal nerve anatomy with accompanying images from the strobe.
Change in volume of injectate in injection laryngoplasty measured by ultrasound compared to amount injected after procedure and at follow-up. | Immediately post-intervention and at 4 week follow-up visit
  The volume will be recorded in mL.
Presence, bulk, and function of tongue, suprahyoid, and infrahyoid musculature on ultrasound for patients with and without swallowing complaints. | Day 1
  This is a qualitative outcome measure. Providers will provide a description of the tongue, suprahyoid, and infrahyoid musculature on ultrasound for patients with and without swallowing complaints.
Evaluation of suprahyoid musculature on ultrasound for patients with muscle tension dysphonia. | Day 1
  This is a qualitative outcome measure. Providers will provide a description of the suprahyoid musculature on ultrasound for patients with muscle tension dysphonia.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Rameau, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No